CLINICAL TRIAL: NCT00003584
Title: A Phase II Trial of Combination Vinorelbine-Estramustine With or Without Prednisone for High Risk and Recurrent, Advanced and Metastatic Renal Cell Carcinoma
Brief Title: Combination Chemotherapy With or Without Prednisone in Treating Patients With Recurrent and/or Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: UNM-1598C; CDR0000066653 (Registry Identifier: PDQ (Physician Data Query)); NCI-V98-1477
Record Dates: First submitted 1999-11-01; First posted 2004-06-09 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Estramustine; Prednisone; Vinorelbine

INTERVENTIONS:
Drug: estramustine phosphate sodium
Drug: prednisone
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Prednisone may help to relieve symptoms in patients with recurrent and/or metastatic kidney cancer.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy consisting of vinorelbine and estramustine with or without prednisone in treating patients who have recurrent and/or metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the response rate of vinorelbine and estramustine in patients with metastatic and/or recurrent renal cell carcinoma. II. Obtain pilot data exploring the value of anti-inflammatory treatment in the management of severe systemic symptoms and improvement of treatment tolerance in this patient population.

OUTLINE: Patients are stratified according to number of risk factors (0,1 versus 2 versus 3). Patients receive vinorelbine IV on days 1, 8, 15, 22, 28, and 35. Patients also receive estramustine orally twice per day on days 1-7 and an increased dose on days 8-42. A tapered dose of oral prednisone is given to patients with an elevated erythrocyte sedimentation rate. A course of treatment consists of 6 weeks of treatment followed by 2 weeks of rest. Patients with stable disease may receive up to 4 courses of treatment. Patients who achieve a partial response may undergo surgical resection followed by up to 2 additional courses of treatment or an interleukin-2 treatment regimen. Patients with a complete response receive 1 additional course of treatment. Patients are followed until death.

PROJECTED ACCRUAL: A maximum of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic and/or recurrent renal cell carcinoma Bidimensionally measurable disease required (outside any prior radiation fields) No untreated brain metastases

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant or nursing Fertile patients must use effective contraception No other serious illness No serious active infection requiring therapy HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic therapy Chemotherapy: No prior vinca alkaloid No other concurrent chemotherapy Endocrine therapy: No concurrent hormone therapy No concurrent corticosteroids (topical or inhaled corticosteroids allowed) Radiotherapy: At least 4 weeks since prior radiotherapy Less than 25% of bone marrow irradiated No concurrent radiotherapy Surgery: At least 3 weeks since prior surgery Other: No other concurrent investigational drugs

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 1998-07; Primary Completion 2000-12 (Actual); Study Completion 2000-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Elias, MD, Study Chair — University of New Mexico Cancer Center
Locations (1):
- University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico, United States